CLINICAL TRIAL: NCT00411203
Title: Double Blind Placebo Controlled Trial of a Protein Kinase C Inhibitor: Tamoxifen Citrate in Treatment of Acute Mania
Brief Title: Tamoxifen in Treatment of Acute Mania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02T-162; AY0001
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Bipolar Disorder
Keywords: Protein kinase C, tamoxifen, acute mania, clinical trial
MeSH Terms: conditions — Bipolar Disorder | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Tamoxifen Citrate (Active Comparator)
  Interventions: Drug: Tamoxifen Citrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamoxifen Citrate
  Arms: Tamoxifen Citrate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Objective: Evidence indicates that the protein kinase C-PKC signaling cascade may be one of the direct targets in treatment of mania. The aim of this study is to investigate whether the PKC inhibitor-tamoxifen has anti-manic properties. Method: Bipolar subjects with manic/mixed episode were randomly assigned to receive either tamoxifen (80mg/day) or identical placebo tablets in 1:1 ratio for three weeks.

DETAILED DESCRIPTION:
Patients aged 18-65 years, diagnosed with Bipolar Disorder (BD), most recent episode manic or mixed, with or without psychotic features were admitted to the inpatient unit at the Dokuz Eylul University, Department of Psychiatry, Izmir, Turkey. Subjects were recruited from the local community, an urban area in the western part of Turkey, surrounding suburbs, and towns as well as all over the country (expert-seeking patients who reached the principle investigator-PI, via the internet and news media) between April, 2003 and June, 2006. All diagnoses were based on the Structured Clinical Interview for the DSM-IV, administered by a trained investigator (AYY). After the protocol explained to the patient and at least one first degree relative, both gave written informed consent for participation of the patient in the trial. The study was approved by the Turkish Ministry of Health, General Directorate of Drugs and Pharmaceutics, Central Review Board, and Local Ethical Committee of Drug Investigations at the Dokuz Eylul University. Subject screening included medical and psychiatric history, physical examination, and laboratory screen including LFTs, TSH, HCG, BUN, Cr, and serum toxicology. All psychotropic medication (except benzodiazepines) was discontinued at least 1 day before randomization. Subjects entering the study were randomly assigned to receive the PKC inhibitor, tamoxifen or identical placebo tablets in a 1:1 ratio and double-blind fashion for 3 weeks. Computer-generated codes were used to create randomization kits (prepared by the ARGEFAR, Izmir, Turkey, a contract research organization). The starting dose of tamoxifen was 20 mg bid. After the first treatment day, daily dose was adjusted upward by 10 mg per day up to 80 mg/d in divided doses. Similar tablet adjustments were applied for the patients in placebo group. Concomitant use of oral lorazepam (2.5mg dissolving tables) was allowed during double-blind therapy as clinically indicated. In cases where lorazepam is thought to be ineffective and the symptoms are such that an antipsychotic is required, risperidone liquid formulations (2-6 mg/day) were used under emergency circumstances. Those subjects who were given risperidone were assumed as drop out at the time of first exposure to risperidone; and new subjects for replacement of those cases have been recruited. Subjects were seen twice daily and investigators (AYY, SG) were on call 24 hours a day.

Assessment tools; Young Mania Rating Scale (YMRS), Hamilton Depression Rating Scale-17 item (HAMD-17), Montgomery-Asberg Depression Rating Scale (MADRS), Clinical Global Impressions-Bipolar Version of Severity of Illness (CGI), and Positive and Negative Syndrome Scale (PANSS) and side effect questionnaire were administered by semi-structured interviews at each week. Vital signs and weight were monitored. The PI, who is trained in the rating instruments and blind to the treatment condition (training and certification at the Massachusetts Hospital, Bipolar Program), performed all the study assessments on a weekly basis by using all the available clinical information, provided by the prospective daily interviews by the investigators, staff reports including the security team' observations, and first degree relative reports.

Power calculations were performed to determine the sample size required to achieve 80% power to detect a difference of 0.40 in the response rate, assuming a 0.15 response rate in placebo using a chi-square test at the .05 level. Assuming 30% drop out and non compliance rate, randomization kits were prepared for 70 subjects. Following eligibility considerations and drop out the final sample size used in the analysis was 50. The primary efficacy variable is defined as the reduction from baseline of the YMRS score after 3 weeks of therapy. Positive treatment response was defined as >=50% decrease in YMRS from baseline to 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of BD I, most recent episode, manic or mixed,
2. ages 18-65,
3. Young Mania Rating Scale (YMRS) score > 20 at screening and baseline,
4. providing written informed consent.

Exclusion Criteria:

1. currently pregnant, planning to become pregnant, or breast feeding,
2. history of any coagulopathies, deep vein thrombosis, pulmonary embolus,
3. a history of hypersensitivity to tamoxifen,
4. drug screen positive for any drug of abuse at screening, active substance abuse in the past 2 weeks or substance dependence in the past 2 months (except nicotine and caffeine),
5. diagnosis of schizophrenia, dementia, delirium, seizure disorder, obsessive compulsive disorder, or major cardiac, hepatic or renal disease that is unstable or that requires medical care,
6. administration of any other investigational drug in the last 30 days,
7. clinically significant suicidal or homicidal ideation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-04; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Reduction from baseline of the Young Mania Rating Scale (YMRS) score | 3 weeks of therapy

SECONDARY OUTCOMES:
Positive treatment response, defined as >= 50% decrease in YMRS | from baseline to 3 weeks
Reduction from baseline of the Clinical Global Impressions-Bipolar Version of Severity of Illness (CGI) score | baseline, 3 weeks of therapy
Reduction from baseline of the Positive and Negative Syndrome Scale (PANSS) score | baseline, 3 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül Yildiz, M.D., Principal Investigator — Dokuz Eylül University, Department of Psychiatry
Locations (1):
- Dokuz Eylül University, Department of Psychiatry, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Kruszewski SP, Paczynski R. Concomitant use of Lorazepam with tamoxifen in bipolar mania clinical trials. Arch Gen Psychiatry. 2009 Jan;66(1):107-8; author reply 108-9. doi: 10.1001/archgenpsychiatry.2008.505. No abstract available. PMID 19124694
- [Result] Yildiz A, Guleryuz S, Ankerst DP, Ongur D, Renshaw PF. Protein kinase C inhibition in the treatment of mania: a double-blind, placebo-controlled trial of tamoxifen. Arch Gen Psychiatry. 2008 Mar;65(3):255-63. doi: 10.1001/archgenpsychiatry.2007.43. PMID 18316672
- [Result] Yildiz A, Vieta E, Leucht S, Baldessarini RJ. Efficacy of antimanic treatments: meta-analysis of randomized, controlled trials. Neuropsychopharmacology. 2011 Jan;36(2):375-89. doi: 10.1038/npp.2010.192. Epub 2010 Oct 27. PMID 20980991
- [Result] Yildiz A, Nikodem M, Vieta E, Correll CU, Baldessarini RJ. A network meta-analysis on comparative efficacy and all-cause discontinuation of antimanic treatments in acute bipolar mania. Psychol Med. 2015 Jan;45(2):299-317. doi: 10.1017/S0033291714001305. Epub 2014 Jul 18. PMID 25036226
- [Derived] Yildiz A, Aydin B, Gokmen N, Yurt A, Cohen B, Keskinoglu P, Ongur D, Renshaw P. Antimanic Treatment With Tamoxifen Affects Brain Chemistry: A Double-Blind, Placebo-Controlled Proton Magnetic Resonance Spectroscopy Study. Biol Psychiatry Cogn Neurosci Neuroimaging. 2016 Mar;1(2):125-131. doi: 10.1016/j.bpsc.2015.12.002. PMID 27231722